CLINICAL TRIAL: NCT04179604
Title: Rationale and Design of a Multicenter Randomized Trial of Levosimendan to Reduce Low Cardiac Output Syndrome in Low Ejection Fraction (≤ 35%) Cardiac Surgery Patients. Spanish Randomized Clinical Trial on Levosimendan (SPARTANS Study)
Brief Title: Spanish Randomized Clinical Trial to Compare Levosimendan Versus Placebo in Postoperative Cardiac Surgery (SPARTANS)
Acronym: SPARTANS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: María de los Ángeles Tena Pajuelo (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry); Canary Foundation (Other); Dr Negrin Hospital Statistician (Unknown); Dr Negrin Hospital Farmacy (Unknown); CRO TRIDE Asesores SL (Unknown); QBE Europe SA/NV (Unknown)
Responsible Party: Sponsor-Investigator, María de los Ángeles Tena Pajuelo, Cardiac Surgeon, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTP-2019-01; 2019-001756-19 (EudraCT Number)
Record Dates: First submitted 2019-11-11; First posted 2019-11-27 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2019-11

CONDITIONS: Cardiac Output, Low
Keywords: Poor left ventricule eyection fraction; Levosimendan; Cardiac surgery; Preoperative Treatment; Low cardiac output syndrome; Clinical Trial
MeSH Terms: conditions — Cardiac Output, Low | interventions — Simendan

STUDY DESIGN:
Intervention Model Description: SPARTANS is a phase II-III, prospective, randomized, triple-blind, placebo-controlled, multicenter clinical trial to evaluate the efficacy of levosimendan in decrease perioperative low cardiac output Syndrome in patients with preoperatively severe left ventricular dysfunction (LVEF ≤ 35%) who will be scheduled for cardiac surgery on cardipulmonary bypass. Follow-up duration will be one year.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Researches will use a computer-generated permuted block randomization established by an independent Statistician. Pharmacy of each hospital will prepare randomized treatment, without being involved in the trial. Patients and physicians will be blind to the randomized therapeutic strategy that each patient will receive. The data will be entered into a specific electronic database in an anonymized and dissociated manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levosimemdam (Experimental): Levosimendan 2.5 mg / ml concentrate for solution for infusion. A 5 ml vial contains 12.5 mg of levosimendan. The concentrate is a clear solution, yellow or orange, for dilution before administration. The study drug infusion will start one day before surgery in an Intensive Care Unit with at least 8 hours of administration before surgery. A continuous infusion at 0.1 µg/kg/min will be administered to complete 24h duration.
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator): Patients in the placebo group will receive a water-soluble vitamin B2 concentrate with 0.4 mg / ml sodium riboflavin phosphate to obtain the same color as the preparation of levosimendan and ethanol anhydrous 100 mg / ml to resemble the levosimendan odor, which will be administered at the same levosimendan infusion rate.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Levosimendan — Levosimendan SIMDAX 2.5 mg / ml concentrate for solution for infusion. The concentrate is a clear solution, yellow or orange, for dilution before administration. A 5 ml vial contains 12.5 mg of levosimendan. The study drug infusion will start one day before surgery in an Intensive Care Unit with at least 8 hours of administration before surgery. A continuous infusion at 0.1 µg/kg/min will be administered to complete 24h duration.
  Other Names: SIMDAX
  Arms: Levosimemdam
Drug: Placebos — Patients in the placebo group will receive a water-soluble vitamin B2 concentrate with 0.4 mg / ml sodium riboflavin phosphate to obtain the same color as the preparation of levosimendan and ethanol anhydrous 100 mg / ml to resemble the levosimendan odor, which will be administered at the same levosimendan infusion rate.
  Arms: Placebo

SUMMARY:
Low cardiac output Syndrome (LCOS) is a complication that appears in approximately 20% of cardiac surgeries with extracorporeal circulation. LCOS is associated with increased mortality, delayed recovery and prolonged hospital stay. The Spanish Randomized Clinical Trial on Levosimendan (brand name: Sindax) (SPARTANS) aims to demonstrate the effectiveness of the preoperative use of Levosimendan in reducing LCOS in patients with poor left ventricle ejection fraction (LVEF) undergoing elective cardiac surgery.

SPARTANS study is a multicenter, randomized triple-blind, placebo-controlled trial. 300 patients with LVEF ≤ 35%, undergoing elective cardiac surgery will be recruited from 9 Spanish hospitals and randomized into two groups: Preoperative administration of levosimendan or placebo for 24 hours. The study drug will be started as a continuous infusion (0.1 µg/kg/min) at least 8 hours before surgery to complete 24h duration.

The primary endpoint will be 30-day LCOS. It will be evaluated using any of the following criteria:

1) postoperated cardiac index ≤2.0 L / min / m2, 2) a need to implant a intra-aortic balloon pump/ left ventricular assist device, 3) a vasoactive inotropic scale (VIS) > 5.5.

The secondary end-point will be composite event rate at one year including any of the following events: death from any cause, need for renal replacement therapy or dialysis and LCOS.

The sample size is based on the assumption that levosimendan reduces LCOS by 50% being necessary a sample size of 300 patients to carry out the study.

The Research Team of each hospital, will carry out the clinical follow-up by telephone or clinical interview of the patient according to the time intervals: 30 days and 1 year. We estimate that the total sample size of 300 patients will be reached in 2-2.5 years.

In conclusion, the effectiveness of levosimendan has not yet been reported with a good evidence in cardiac surgery. The purpose of the "Spanish Randomized Clinical Trial on Sindax" (SPARTANS) trial is to evaluate the beneficial effect of preoperative use of levosimendan compared with placebo to reduce perioperative LCOS in patients undergoing cardiac surgery with poor LVEF ≤ 35%.

DETAILED DESCRIPTION:
Low cardiac output syndrome (LCOS) is defined, by the Working Group of Cardiac Intensive Care of the Spanish Society of Intensive, Critical Medicine and Coronary Units, as a cardiac index (CI) <2.2 l / min / m2. LCOS is due to left and/or right ventricular failure and may be associated with pulmonary congestion and may occur with normal or low blood pressure. LCO after cardiac surgery is associated with increased mortality, delayed functional and organic recovery and prolonged stay in the Intensive Care Unit. It is characterized by a decrease in cardiac function, a reduction in oxygen supply and subsequent tissue hypoxia, together with signs of tissue hypoperfusion (peripheral coldness, confusion, oliguria and elevated lactate level) and in absence of hypovolemia.

LCOS appears in approximately 20% of cardiopulmonary bypass (CPB) surgeries. Levosimendan, a calcium-sensitizing inotrope and an ATP-sensitive potassium channel opener, has been reported to be effective in decreasing LCOS and mortality after cardiac surgery. Simdax, which is its trade name, is indicated for the short-term treatment of severe acute decompensation of chronic heart failure in situations where conventional treatment is not sufficient or in cases where an inotropic support is considered appropriate.

The recent publication of 2 large randomized clinical trials LEVO-CTS and LICORN failed to meet any benefit of levosimendan in terms of survival in cardiac surgery. Still, in a recently published meta-analysis, researchers showed that Levosimendan is effective in reducing low-cardiac output Syndrome compared to placebo (14.8% in the Levosimendan group versus 29.0% in the placebo group; RR = 0.40 , 95% CI = 0.22-0.73; P = 0.003).

The purpose of the "Spanish Randomized Clinical Trial on Sindax" (SPARTANS) trial is to evaluate the beneficial effect of preoperative use of Levosimendan compared with placebo to reduce perioperative LCOS in patients undergoing cardiac surgery with poor LVF.

The study was approved by the Ethical Committee of all participating centers. SPARTANS is a phase III, randomized, triple-blind, placebo-controlled, multicenter clinical trial to evaluate the efficacy of levosimendan in decrease perioperative LCOS in patients with preoperatively severe left ventricular dysfunction (LVEF ≤ 35%) who will be scheduled for cardiac surgery on CBP.

The sample size was calculated based on an earlier meta-analysis (Tena MA, Urso S et al. Levosimendan versus placebo in cardiac surgery: a systematic review and a meta-analysis. Interact Cardiovasc Thorac Surg. 2018 27: 677-685) where researches document that Levosimendan is effective in reducing the rate of low postoperative cardiac output Syndrome compared to placebo (14.8% in the Levosimendan group versus 29.0% in the placebo group; RR = 0.40, 95% CI = 0.22-0.73; P = 0.003 ). Thus, considering a type I error of 0.05, a type II error of 0.20, a ratio of 1/1, an event rate of 29% in the Placebo group and an event rate of 15% in the Levosimendan group, a sample population of at least 137 patients for each group is required. Assuming a 9,5% patient drop rate, researches obtain a total sample of 300 patients (MedCalc Software bvba, Ostende, Belgium, http://www.medcalc.org, 2017).

Thus, 300 patients will be enroll at 9 Spanish University hospitals scheduled for isolated aortic valve replacement (AVR) and/or coronary artery bypass grafting (CABG) with cardiopulmonary bypass (CPB). All enrolled patients will have a preoperative LVEF equal to, or less than 35 % detected by echocardiography measurement one week before surgery and will be required to give written informed consent, prior to being properly informed about participation in the trial, before enrollment. Researches hope to recruit 300 patients in 2 years.

150 patients will receive randomly levosimendan and another 150 patients placebo with identical appearance and doses to the medication under study. The study drug or placebo infusion will start one day before surgery in an Intensive Care Unit with at least 8 hours of administration before surgery. A continuous infusion at 0.1 µg/kg/min will be administered to complete 24h duration. If patients once randomized, suffering from one adverse event during the infusion, they will be registered stopping the infusion. In the case that the adverse event occurred in the postoperative period and if it was demonstrated due to the cause of the medication under study, it will be registered too.

Researches will use a computer-generated permuted block randomization established by an independent statistician. Pharmacy of each hospital will prepare randomized treatment, without being involved in the trial. Patients and physicians will be blind to the randomized therapeutic strategy that each patient will receive. The data will be entered into a specific electronic database in an anonymized and dissociated manner.

Patients Data will be collected by a Research Team for each participating hospital that will consist of at least one Cardiac Surgeon, an Anesthesiologist and a specialist in postoperative Critical Care. These investigators will receive training about patient selection and clinical events registration with the help of Contract Research Organization (CRO TRIDE ASESORES SL). This CRO will carry out regulatory execution of the trial, oversight and collection of electronic data, follow up and scientific regulation of procedures between different ethical Committees and hospitals involved. All data will be evaluated by trial main researcher and CRO identifying possible data collection errors and acting according to good clinical practice. The identification of a clinical event will be done by absolute majority by the members of the Research Team.

Anesthesia, surgery and CBP will be performed according to standard operating procedures and following the usual clinical practice of each hospital.

The primary endpoint is to demonstrate that preoperative levosimendan administration in patients undergoing AVR and/or CABG with poor LVEF ≤ 35% halve perioperative LCOS during the first 30 days of surgery. The secondary endopoint is to analyze composite event rate up to one year after surgery. The results will be expressed as means (±SD) or as medians and interquartile range to express quantitative variables. Qualitative variables will be expressed by frequency and percentage. Categorical variables will be compared by Fisher's exact test and continuous variables will be compared by Student's test or Mann-Whitney U. Incidence of composite endpoint will be compared between the two groups using a Chi-square test o Fisher's exact test. The Friedman or Anova test of repeated measures will be used to compare measures repeated through the study time. The risk factors will be expressed through relative risks (ratio of cumulative incidents), Odds Ratio or Hazard Ratio and their respective confidence intervals. Survival curves will be compared using the Log-rank test. All analyzes will be performed 2-sided and with an alpha level of 5%. All analyzes will be performed using the R program, version 3.5.2 or higher (R Foundation). The statistical calculation procedure will be carried out by an independent statistician and during the third year.

Researches will follow the recommendations of Helsinki and Consort to carry out the trial and give greater validity to study results.The patients, sponsor or researchers included in trial will not receive financial compensation and declare that there has been no conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written informed consent
* LVEF ≤35% detected by echocardiography carried out at least one week before surgery.
* Scheduled AVR or/and Scheduled CABG with CBP.

Exclusion Criteria:

* Previous levosimendan administration.
* Emergency operation.
* Kidney or liver trasplant or awaiting it.
* Hepatic cirrhosis Child C. In case Child B, contact coordinating center.
* Any degree of preoperative right ventricular failure.
* Preoperative creatinine > 2 mg / dl.
* Valve desease other than aortic.
* Renal failure requering dialysis (or creatinine clearance < 30ml / min).
* Hemodynamic instability (need for inotropics, unstable angina, acute myocardial infarction, intra-aortic balloon pump).
* Patients underwent previous cardiac surgery.
* Allergy or hypersensitivity to levosimendan or any of its excipients
* Severe hypotension (sistolic arterial tension < 80 mmHg or mean arterial pressure <50 mmHg ) and tachycardia ( heart rate >130 bpm).
* History of Torsades de Pointes.
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with LCOS | up to 30 days of cardiac surgery
  LCOS will be considered if:
  1) Postoperated cardiac index ≤2.0 L / min / m2 (liters / minute / square meter)
Number of Participants with LCOS | up to 30 days of cardiac surgery
  LCOS will be considered if:
  2) The need to implant an intra-aortic balloon pump
Number of Participants with LCOS | up to 30 days of cardiac surgery
  LCOS will be considered if:
  3) The need to implant a left ventricular assistance device
Number of Participants with LCOS | up to 30 days of cardiac surgery
  LCOS will be considered if:
  4) To have a vasoactive inotropic scale (VIS) > 5.5 Vasoactive inotropic scale will be measured following the following formula: inotropic scale (IS) + 10 x Milrinone (μg / kg / min) + 100 x norepinephrine (μg / kg / min) + 10000 × vasopressin (U / kg / min).
  The inotropic scale (SI) will be calculated using the following formula: Dopamine (μg / kg / min) + Dobutamine (μg / kg / min) + 100 × adrenaline (μg / kg / min).

SECONDARY OUTCOMES:
Composite event rate | up to one year after surgery
  includes the following options:
  1) Death from any cause (proportion of patients with mortality from any case in each group Levo versus Placebo)
Composite event rate | up to one year after surgery
  includes the following options: 2) The need for renal replacement therapy or dialysis (proportion of patients in each group Levo versus Placebo)
Composite event rate | up to one year after surgery
  includes the following options: 3) LCOS (proportion of patients in each group Levo versus Placebo) It is calculated by adding the proportions of each of the 3 events described above.

OTHER OUTCOMES:
Number of Patients with need for renal replacement therapy or dialysis | up to 30 days
  Need for renal replacement therapy or dialysis in each group
Intensive Care Unit stay | until discharge from Intensive Care Unit
  days in Intensive Care Unit Stay (calculate the average days of stay of all patients in each levo and placebo group)
Total post-surgical stay | until discharge from hospital
  days from surgery to hospital discharge (arithmetic average)
Number of Patients with hospital cardiac mortality | until discharge from hospital
  Hospital cardiac mortality
Number of Patients with need for ventricular assistance or intra-aortic balloon pump | up to 1 year after surgery
  Need for ventricular assistance or intra-aortic balloon in each group

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ángeles T Tena Pajuelo, Cardiac surgery, Principal Investigator — Doctor Negrin University Hospital; Marta P Perez de Lis Novo, anesthesiology, Principal Investigator — A Coruña University Complex; Juan B Bustamante Munguira, Cardiac surgery, Principal Investigator — Valladolid UNIVERSITY CLINICAL HOSPITAL; Marc V Vives Santacana, anesthesiology, Principal Investigator — Doctor Joseh Trueta, Girona university clinical Hospital; Elisabet B Berastegui Garcia, Cardiac surgery, Principal Investigator — GERMANS TRIAS I PUJOL DE BADALONA University Hospital; Pedro M Muñoz Ramirez, anesthesiology, Principal Investigator — 12 de Octubre University Hospital; Ana Isabel G Gonzalez Roman, anesthesiology, Principal Investigator — Puerta del Hierro University Hospital; Gemma S Sanchez Espin, Cardiac Surgery, Principal Investigator — Virgen de la Victoria University Hospital; Emiliano Andres R Rodriguez Caulo, Cardiac Surgery, Principal Investigator — Virgen Macarena University Hospital
Locations (9):
- Spain (9):
  - GERMANS TRIAS I PUJOL DE BADALONA university Hospital, Badalona, Barcelona
  - Doctor Josep Trueta university Hospital, Girona, Gerona
  - Doctor Negrin University Hospital, Las Palmas de Gran Canaria, Gran Canarias
  - Puerta del Hierro University Hospital, Majadahonda, Madrid
  - Virgen de la Victoria University Hospital, Málaga, Malaga
  - A coruña UNIVERSITY HOSPITAL COMPLEX A CORUÑA, A Coruña
  - 12 de Octubre University Hospital, Madrid
  - Virgen Macarena University Hospital, Seville
  - Valladolid universitary Hospital, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Once the statistical analysis is completed during third year, the results of the study will be presented at the Congresses of the Spanish Society of Cardiothoracic Surgery. The informs and conclusions obtained by the statistical analysis of the study population will be sent for publication in impact journals. We will share all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From the fourth year of the study and they will be available indefinitely where it is published.

REFERENCES:
- [Result] Tena MA, Urso S, Gonzalez JM, Santana L, Sadaba R, Juarez P, Gonzalez L, Portela F. Levosimendan versus placebo in cardiac surgery: a systematic review and meta-analysis. Interact Cardiovasc Thorac Surg. 2018 Nov 1;27(5):677-685. doi: 10.1093/icvts/ivy133. PMID 29718383
- [Result] Landoni G, Mizzi A, Biondi-Zoccai G, Bruno G, Bignami E, Corno L, Zambon M, Gerli C, Zangrillo A. Reducing mortality in cardiac surgery with levosimendan: a meta-analysis of randomized controlled trials. J Cardiothorac Vasc Anesth. 2010 Feb;24(1):51-7. doi: 10.1053/j.jvca.2009.05.031. Epub 2009 Aug 22. PMID 19700350
- [Result] Niu ZZ, Wu SM, Sun WY, Hou WM, Chi YF. Perioperative levosimendan therapy is associated with a lower incidence of acute kidney injury after cardiac surgery: a meta-analysis. J Cardiovasc Pharmacol. 2014 Feb;63(2):107-12. doi: 10.1097/FJC.0000000000000028. PMID 24126568
- [Result] Levin R, Degrange M, Del Mazo C, Tanus E, Porcile R. Preoperative levosimendan decreases mortality and the development of low cardiac output in high-risk patients with severe left ventricular dysfunction undergoing coronary artery bypass grafting with cardiopulmonary bypass. Exp Clin Cardiol. 2012 Sep;17(3):125-30. PMID 23620700